CLINICAL TRIAL: NCT03083301
Title: Cardiac Resynchronization Therapy: Relevance of the Surgical Approach in the Implantation of the Left Ventricular Probe
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, CHU Brugmann, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-cardiac resynchronization
Record Dates: First submitted 2017-03-08; First posted 2017-03-20 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cardiac Insufficiency
Keywords: Cardiac resynchronisation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac insufficiency: Patients with cardiac insufficiency (i.e in NYHA class III or IV) or refractory to optimal medical treatment (155 patients since 2003) in the Brugmann University Hospital, in the cardiac surgery department
  Interventions: Other: Medical Files data extraction

INTERVENTIONS:
Other: Medical Files data extraction — Medical Files data extraction

SUMMARY:
Heart failure is very common and reaches more than 56 million people worldwide. 17 to 45 percent die in the first year of hospitalization. The most affected populations live in Western countries like Europe or the USA.

It is defined by a set of signs and symptoms such as dyspnea, asthenia, edema or tachycardia but must be objectified, preferably by ultrasound. Its basic treatment is based on a lifestyle improvement and a reduction of the risk factors (hypertension, dyslipidemia, diabetes, ...), as well as an optimal medical treatment based on ACE inhibitors, B-blockers, ARA2 (Sartans), spironolactone or digoxin.

When the optimal treatment is no longer working and that the cardiac desynchronization is demonstrated, be it atrio-ventricular, inter-ventricular or intra-ventricular, the patient can benefit from a three-probes cardiac resynchronization to resynchronize the two ventricles. The classic approach, performed by a cardiologist, is to perform an endovenous procedure in order to place the 3 probes under local anesthesia.The first one goes in the right atrium, the second one in the right ventricle and the third one goes in the left ventricle. It is the placement of this third one that often causes trouble. It is more difficult to place since it must pass through the coronary sinus, outside of the heart, unlike the first two probes that are placed endocavitary. When the practitioner fails to place the probe correctly or obtains inappropriate levels of detection, stimulation, or impedance thresholds, a cardiac surgeon must intervene and carry out a mini-thoracotomy.

The CHU Brugmann Hospital is in favor of a mixed surgical approach. The probes are placed by a cardiac surgeon, who first starts by a endo-venous placement under local anesthesia. If that approach fails, the local anesthesia can be transformed into general anesthesia at the same operative time and a mini-thoracotomy is performed.

The aim of this study is to evaluate the immediate impact of this surgical management within the CHU Brugmann hospital, in patients suffering from cardiac insufficiency despite proper medication.The hypothesis is that the mixed surgical approach improves the prognosis of cardiac resynchronization.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent cardiac resynchronization within the Brugmann University Hospital from 2003 til July 2016
* Cardiac insufficiency, whatever the origin, demonstrated by a cardiologist with demonstrated ventricular asynchronism.

  * With left ventricular ejection fraction <35%
  * And / or a left ventricular diastolic diastolic diameter> 55 mm
  * And / or QRS measuring> 130 milli sec
  * And / or left branch block
* Redo procedure on a pacemaker

Exclusion Criteria:

• Change of case on a patient who has already benefited from a triple chamber stimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiac insufficiency (i.e in NYHA class III or IV) or refractory to optimal medical treatment (155 patients since 2003) in the Brugmann University Hospital, in the cardiac surgery department.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Direct failure rate of the mixed approach | 7 years
  Direct failure rate of the mixed approach
Demographic data | 7 years
  Demographic data (descriptive analysis)
Risks factors | 7 years
  Descriptive analysis of the risks factors linked to the failure of the procedure
Type of cardiopathy | 7 years
  Type of cardiopathy
PR interval | 7 years
  PR interval
QRS interval | 7 years
  QRS interval

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wauthy, MD, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No